CLINICAL TRIAL: NCT06828159
Title: Effects of Dietary Wild Blueberries on Gut Health and Inflammation and Joint Pain
Brief Title: Dietary Wild Blueberries and Joint Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Oklahoma Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: OMRF WB01; WBANA01 (Other Grant/Funding Number: WBANA)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: Gut -Microbiota; Inflammation Biomarkers; Pain Assessment; Joint Pain
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wild blueberries (Experimental): 25g freeze-dried wild blueberries daily for 12 weeks
  Interventions: Dietary Supplement: Wild blueberry
- Placebo (Placebo Comparator): Placebo powder free from polyphenols matched for calories
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wild blueberry — Freeze-dried wild blueberry powder 25g/day
  Arms: Wild blueberries
Dietary Supplement: Placebo — Placebo powder matched for calories and no polyphenols
  Arms: Placebo

SUMMARY:
The goal of this proposed study is to examine the effects of dietary wild blueberries on gut microbiome, serum markers of inflammation, and joint function in adults. Each participant will consume 25g freeze-dried blueberries or matched placebo powder for 12 weeks, with a 2-week washout phase between.

ELIGIBILITY:
Inclusion Criteria:

* Adults with documented multi-joint/knee arthritis

Exclusion Criteria:

* inability to give informed consent
* pregnancy or lactation
* planned knee replacement surgery
* allergy or contraindication to berries
* recent trauma of the knee responsible of the symptomatic knee
* intra-articular injection in the target knee/hip in the last 3 months
* oral corticosteroid therapy ≥ 5 mg/day (prednisone equivalent) at baseline
* use of berry extracts in the last 3 months
* special diets
* cancer treatment
* bone diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Serum biomarkers of joint function | 12 weeks
  Serum biomarkers of inflammation and cartilage degradation will be measured in the wild blueberry and placebo groups and compared for outcomes. Pain scores will also be measured using self-reported questionnaires.

SECONDARY OUTCOMES:
Gut microbiome | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- OMRF, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No